CLINICAL TRIAL: NCT04861701
Title: Effect and Predictors for Hot Flush in Women Undergoing Static Stretching Exercise : A Randomized Controlled Trial
Brief Title: Effect and Predictors for Hot Flush in Women Undergoing Static Stretching Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Mei-Wun Tsai, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: YM109101E
Record Dates: First submitted 2021-04-26; First posted 2021-04-27 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching exercise group (SE) (Experimental): All subjects will be assigned to the experimental or control group by randomization. Thus, there will be totally 2 groups : Stretching exercise group (SE) and Control group (CON).
  Interventions: Behavioral: Static stretching exercise
- Control group (CON) (No Intervention): All subjects will be assigned to the experimental or control group by randomization. Thus, there will be totally 2 groups : Stretching exercise group (SE) and Control group (CON).

INTERVENTIONS:
Behavioral: Static stretching exercise — The intervention of this study is home-based stretching exercise. The experimental group will receive 6 stretching exercises which stretch 60 seconds for each side (left or right) of each movement, and relax for 10-20 seconds between the movements. It will take 10-15 minutes every day for continuous 4 weeks. The 6 stretching exercises include : (1) pectoral muscles + calf muscles ; (2) quadriceps ; (3) levator scapulae ; (4) gluteal muscles ; (5) hamstrings ; (6) trunk side-flexors.
  Arms: Stretching exercise group (SE)

SUMMARY:
This study investigates the effect and predictors of static stretching exercise on hot flush in women after performing 4-week stretching exercises.

DETAILED DESCRIPTION:
Hot flush (HF) is the most common symptom among menopausal syndrome and can significantly affect women's quality of life. Considering the risk of hormone therapy, the behavioral therapies have been proposed for the alternative treatment of HF. However, the exercise prescription for women with HF is controversial. Previous studies show the inconsistent effect of aerobic exercise on HF, and a moderate-to-high intensity exercise seems to aggravate HF frequency and severity. Recent studies have shown that static stretching exercise could improve HF in middle-aged women, but the related research is quite few, and the physiological mechanism as well as predictors for responders who can benefit from stretching exercise are still not clear. The knowledge of predictors for responders will provide clinicians and clients with HF symptoms to choose static stretching exercise as their treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-65 years old.
2. With hot flashes.
3. No current therapies such as hormone therapy, psychotropic medications, or sleeping pills for the past 6 months.
4. With ability to follow instructions of stretching exercise.

Exclusion Criteria:

1. SBP >160 mmHg or DBP >100 mmHg
2. Medical condition under investigation or unstable condition that could affect hot flashes, like thyroid disease.
3. Any medical condition limiting the ability to participate the exercise.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with hot flashes
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Hot flush frequency | pre-intervention
  Frequency of hot flush (time/day)
Hot flush frequency | week 1 of intervention period
  Frequency of hot flush (time/day)
Hot flush frequency | week 2 of intervention period
  Frequency of hot flush (time/day)
Hot flush frequency | week 3 of intervention period
  Frequency of hot flush (time/day)
Hot flush frequency | week 4 of intervention period (post-intervention)
  Frequency of hot flush (time/day)
Hot flush score | pre-intervention
  The sum of mean hot flushes multiplied by severity (mild x 1, moderate x 2, severe x 3)
Hot flush score | week 1 of intervention period
  The sum of mean hot flushes multiplied by severity (mild x 1, moderate x 2, severe x 3)
Hot flush score | week 2 of intervention period
  The sum of mean hot flushes multiplied by severity (mild x 1, moderate x 2, severe x 3)
Hot flush score | week 3 of intervention period
  The sum of mean hot flushes multiplied by severity (mild x 1, moderate x 2, severe x 3)
Hot flush score | week 4 of intervention period (post-intervention)
  The sum of mean hot flushes multiplied by severity (mild x 1, moderate x 2, severe x 3)

SECONDARY OUTCOMES:
Standard deviation of NN intervals (SDNN) | pre-intervention
  SDNN represents total heart rate variability. (unit: ms)
Standard deviation of NN intervals (SDNN) | week 4 of intervention period (post-intervention)
  SDNN represents total heart rate variability. (unit: ms)
Absolute total power | pre-intervention
  Absolute total power represents total activity of autonomic nervous system. (unit: ms^2)
Absolute total power | week 4 of intervention period (post-intervention)
  Absolute total power represents total activity of autonomic nervous system. (unit: ms^2)
Low frequency in normalized unit (LF norm) | pre-intervention
  LF norm represents sympathetic nerve activity.
Low frequency in normalized unit (LF norm) | week 4 of intervention period (post-intervention)
  LF norm represents sympathetic nerve activity.
High frequency in normalized unit (HF norm) | pre-intervention
  HF norm represents parasympathetic nerve activity.
High frequency in normalized unit (HF norm) | week 4 of intervention period (post-intervention)
  HF norm represents parasympathetic nerve activity.
Percentage of low frequency (LF%) | pre-intervention
  LF% represents sympathetic nerve activity.
Percentage of low frequency (LF%) | week 4 of intervention period (post-intervention)
  LF% represents sympathetic nerve activity.
Percentage of high frequency (HF%) | pre-intervention
  HF% represents parasympathetic nerve activity.
Percentage of high frequency (HF%) | week 4 of intervention period (post-intervention)
  HF% represents parasympathetic nerve activity.
LF/HF ratio (L/H ratio) | pre-intervention
  L/H ratio represents autonomic nerve balance.
LF/HF ratio (L/H ratio) | week 4 of intervention period (post-intervention)
  L/H ratio represents autonomic nerve balance.
Muscle flexibility of upper extremities | pre-intervention
  Apley's scratch test (unit: cm)
Muscle flexibility of upper extremities | week 4 of intervention period (post-intervention)
  Apley's scratch test (unit: cm)
Muscle flexibility of lower extremities | pre-intervention
  Sit-and-reach test (unit: cm)
Muscle flexibility of lower extremities | week 4 of intervention period (post-intervention)
  Sit-and-reach test (unit: cm)
Vascular endothelial function | pre-intervention
  Reflective index (RI) (unit：％)
Vascular endothelial function | week 4 of intervention period (post-intervention)
  Reflective index (RI) (unit：％)
Hot Flush Related Daily Interference Scale (HFRDIS) | pre-intervention
  Hot Flush Related Daily Interference Scale (HFRDIS), minimum value : 0, maximum value : 100, higher scores mean a worse outcome
Hot Flush Related Daily Interference Scale (HFRDIS) | week 4 of intervention period (post-intervention)
  Hot Flush Related Daily Interference Scale (HFRDIS), minimum value : 0, maximum value : 100, higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: I-Hsuan Lu, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming University, Taipei, Taiwan